CLINICAL TRIAL: NCT01920386
Title: A Randomized, Double-blind, Active-controlled, Parallel, Multicenter Phase 3 Study of Tramadol Hydrochloride/Acetaminophen SR Tab. & Tramadol Hydrochloride/Acetaminophen Tab. in Acute Toothache Patients After Teeth Extraction Surgery
Brief Title: Phase 3 Study of Tramadol Hydrochloride/Acetaminophen SR Tab. & Tramadol Hydrochloride/Acetaminophen Tab. in Acute Toothache Patients After Teeth Extraction Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW 0919 302 Version 1.0
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Acute Toothache Patients Above Moderate Pain After Teeth Extraction Surgery
Keywords: Acute Toothache; Wontran; Wontran SR Tab.; Tramadol Hydrochloride/Acetaminophen
MeSH Terms: interventions — Tramadol; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Tramadol hydrochloride/Acetaminophen Tab. (Active Comparator): 1tab PO within 5hours from teeth extraction
  Interventions: Drug: Tramadol hydrochloride/Acetaminophen Tab.
- Tramadol hydrochloride/Acetaminophen SR Tab. (Experimental): 1tab PO within 5hours from teeth extraction and then 1tab more after 6hours
  Interventions: Drug: Tramadol hydrochloride/Acetaminophen SR Tab.

INTERVENTIONS:
Drug: Tramadol hydrochloride/Acetaminophen Tab.
  Arms: Tramadol hydrochloride/Acetaminophen Tab.
Drug: Tramadol hydrochloride/Acetaminophen SR Tab.
  Arms: Tramadol hydrochloride/Acetaminophen SR Tab.

SUMMARY:
A randomized, double-blind, active-controlled, parallel, multicenter Phase 3 study of Tramadol hydrochloride/Acetaminophen SR Tab. & Tramadol hydrochloride/Acetaminophen Tab. in Acute Toothache Patients above Moderate Pain after Teeth Extraction Surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males/Females aged over 20 years
2. Patients with over 2 impacted wisdom teeth in the upper and lower jaws
3. Pain VAS Value over 50 mm evaluated as 100mm VAS
4. Subjects who voluntarily or legal guardian agreed with written consent

Exclusion Criteria:

1. Patients with severe heart disease, uncontrol hypertension, diabetes
2. Patients who had taken a long period NSAID (eg. celecoxib, rofecoxib naproxen etc) within 3 days from the screening point
3. Patients who had taken short-time anesthetic drugs and analgesics within 12 hours from the screening point (except short-time anesthetics before or during surgery)
4. Patients with aspirin asthma(asthma seizure caused by NSAIDs) or medical history
5. Patients with severe respiratory depression

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
SPID ; Sum of the pain intensity differences | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12 hour